CLINICAL TRIAL: NCT00549328
Title: A Phase II, Non-randomized, Multi-center Study to Evaluate the Efficacy and Safety of Pazopanib (GW786034) in Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: Monotherapy Pazopanib in Subjects With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study enrolment was delayed in starting and too slow to support further development in this setting
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 109609
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: anti-angiogenesis; Non-small cell lung cancer,; pazopanib (GW786034)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pazopanib

ARMS (1):
- Pazopanib Open-label (Experimental): Single-arm, non-randomised, single-stage pazopanib monotherapy.
  Interventions: Drug: Pazopanib (GW786034)

INTERVENTIONS:
Drug: Pazopanib (GW786034) — Pazopanib monotherapy

SUMMARY:
This study is designed to evaluate the efficacy and safety of monotherapy pazopanib (a small molecule tyrosine kinase inhibitor of VEGFR-1, VEGFR-2, VEGFR-3, PDGF, and c-kit) in subjects with advanced (Stage IIIB or IV) non-small cell lung cancer.

DETAILED DESCRIPTION:
Study 109609 is a single-arm, non-randomized, single-stage Phase II study of pazopanib in subjects with Stage IIIB or IV non-small cell lung cancer who have progressed after one or two prior regimens of systemic therapy. The study will be conducted at a limited number of institutions in the US. A total of 40 evaluable subjects will be enrolled and treated. Pazopanib will be given at a dose of 800mg (as determined by previous Phase I studies) orally once per day. Subjects may continue to receive study drug for up to two years unless they experience disease progression or withdraw from treatment for other reasons, or unless the Sponsor terminates the study. A rollover study may be available to those subjects who are exhibiting clinical benefit (stable disease or better). Evaluable subjects will be assessed for response as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Histologically- or cytologically confirmed diagnosis of Stage IIIB or IV non-small cell lung cancer.
* Failed no more than two prior chemotherapy regimens for Stage IIIB or IV non-small cell lung cancer, including a platinum-containing regimen.
* Brain metastases permitted if subject has been treated with surgery and/or radiation therapy more than 4 weeks prior to date of first dose and is stable for at least one week off steroids.
* 18 years of age or older.
* Eastern Cooperative Oncology Group performance status of at least 2.
* Measurable disease according to RECIST.
* Adequate organ system function.
* Females may be eligible to enroll if they are of non-childbearing potential (surgically sterile or post-menopausal)or are using appropriate contraception methods.

Exclusion Criteria:

* Prior malignancy - unless disease-free for at least 3 years, or have had completely resected non-melanomatous skin cancer or successfully treated in situ carcinoma.
* History or clinical evidence of central nervous system metastases or leptomeningeal carcinomatosis, except for subjects with previously-treated CNS metastases, who are asymptomatic, and have had no requirement for steroids or anti-seizure medication for one week prior to first dose of study drug.
* Clinically significant gastrointestinal abnormalities.
* Presence of uncontrolled infection.
* Corrected QT interval greater than 480 msec.
* History of significant cardiovascular condition(s).
* Poorly controlled hypertension (systolic blood pressure of 140mmHG or greater or diastolic blood pressure of 90mmHg or greater).
* History of cerebrovascular accident, pulmonary embolism, or insufficiently treated deep venous thrombosis within the past 6 months prior to first dose of study drug.
* Major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Active bleeding or diathesis.
* Hemoptysis in excess of 2.5mL within 8 weeks of first dose of study drug.
* Serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance with study procedures.
* Use of prohibited medications as defined in protocol.
* Use of an investigational agent, including an investigational anti-cancer agent within 28 days, or 5 half-lives, whichever is longer, prior to first dose of study drug.
* Prior use of any investigational or licensed anti-angiogenic agent, including thalidomide and agents that target platelet-derived growth factor. Prior treatment with bevacizumab or epidermal growth factor receptor tyrosine kinase inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (13):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Duluth, Minnesota
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Sayre, Pennsylvania
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib 800 mg: Pazopanib 800 milligrams (mg) monotherapy given orally once daily
Period: Overall Study
Arm/Group | Pazopanib 800 mg
Started | 14
Completed | 0
Not Completed | 14
Not completed — Adverse Event | 2
Not completed — Disease Progression | 10
Not completed — Death | 1
Not completed — Use of Prohibited Medication | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  White | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Either a Confirmed Complete Response or Partial Response Per RECIST Criteria
Description: The best overall response using Response Evaluation Criteria In Solid Tumors (RESIST) was measured. Complete response is defined as the disappearance of all known lesion(s), confirmed at 4 weeks, and partial response is defined as at least a 30% decrease in the sum of the longest diameters of target lesions taken as a reference to baseline sum of the longest diameters, confirmed at 4 weeks. No formal efficacy analyses were performed due to early termination of the study.
Time Frame: Baseline through End of Study (up to 2 years)
Population: All Treated Population: all participants who met inclusion criteria and willingly consented to participate in the study
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants Who Had a Complete or Partial Response, or Stable Disease
Description: Disease control was measured. Stable disease (SD) is defined as neither partial response (at least a 30% decrease in the sum of the longest diameters of target lesions taken as a reference to baseline sum of the longest diameters, confirmed at 4 weeks) nor progressive disease (PD; a 20% increase in the sum of the longest diameters of target lesions, taken as a reference the smallest sum of the longest diameter recorded since the treatment started or the appearance of one or more new lesions. No formal efficacy analyses were performed due to early termination of the study.
Time Frame: Baseline through End of Study (up to 2 years)
Population: All Treated Population
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival is defined as the interval between the start of treatment and the earliest date of disease progression or death due to any cause, whichever occurs first. No formal efficacy analyses were performed due to early termination of the study.
Time Frame: Baseline through End of Study (up to 2 years)
Population: All Treated Population
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the start of treatment until death due to any cause. No formal efficacy analyses were performed due to early termination of the study.
Time Frame: Baseline through End of Study (up to 2 years)
Population: All Treated Population
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Levels of Circulating Biomarkers in Plasma
Description: Biomarkers are proteins that respond in a unique way to treatment with the study drug; however, levels of proteins were not collected for this measurement. No formal efficacy analyses were performed due to early termination of the study.
Time Frame: Baseline through End of Study (up to 2 years)
Population: All Treated Population
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 0

6. Secondary Outcome: Characterization of Participant Populations by Identification of Intra-tumoral Biomarkers
Description: as for outcome 5
Time Frame: Baseline through End of Study (up to 2 years)
Population: All Treated Population
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Pazopanib 800 mg
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=14)
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=14)
Fatigue (General disorders) | 8
Diarrhea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Stomatitis (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Hair color changes (Skin and subcutaneous tissue disorders) | 3
Weight decreased (Investigations) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.